CLINICAL TRIAL: NCT06249204
Title: Organization-Wide Coaching Intervention of Dementia Care Practice Recommendations: A Cluster Randomized-Control Trial
Brief Title: Patient-Centered Dementia Care Practice Coaching Intervention
Acronym: DCPR_CC3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alzheimer's Disease and Related Disorders Association, Inc (Other)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CC3 - OH_Phase_3
Record Dates: First submitted 2024-01-11; First posted 2024-02-08 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Dementia; Alzheimer Disease
Keywords: person-centered care; dementia care practice recommendations; coaching
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: The study design is a cluster, randomized, no blinded, controlled study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coaching Group (Active Comparator): The intervention group will be exposed to six coaching sessions (one a month for 6 months) as well as a nine month touch point to complete the 3-month post survey. This group will have access to a care community coach, resources and use these supports to create action steps towards adopting and implementing person-centered best practices based on an initial self-assessment of their current practices.
  Interventions: Behavioral: Coaching Group
- Training Group (No Intervention): This group will complete the same pre, immediate post and 3-month post surveys as the intervention group but will receive no intervention during the six month period.

INTERVENTIONS:
Behavioral: Coaching Group — Over a six-month coaching program period, staff members from care communities work with a coach to assess their current level of adoption of Dementia Care Practice Recommendations (DCPR) (published recommendations by Alzheimer's Association) and prioritize areas of need /focus. Teams meet with the coach virtually or in person for 1 hour each month during the six months. Through an action planning and implementation process, care communities are guided to make organization-wide, measurable changes in the areas of (1) policies and procedures, (2) education and training, and/or (3) care practices to increase and maintain person-centered care practices as outlined in the DCPR. Coaches provide ongoing support to the care community through telephone and email support between meetings.
  Other Names: Organization-Wide Coaching Intervention
  Arms: Coaching Group

SUMMARY:
The goal of this clinical trial is to compare staff outcomes in long-term care communities who participate in the intervention versus those who do not. The main questions it aims to answer are: 1. Is employee satisfaction impacted by the intervention and 2. Is dementia care confidence impacted by the intervention. Participants will include monthly coaching visits for the intervention group and completion of surveys pre, immediately post and three-months post. Researchers will compare the intervention group to the control group to see if the intervention impacted the outcomes.

DETAILED DESCRIPTION:
Over a six-month coaching program period, staff members from care communities work with a coach to assess their current level of adoption of Dementia Care Practice Recommendations (DCPR) (published recommendations by Alzheimer's Association) and prioritize areas of need /focus. Teams meet with the coach virtually or in person for 1 hour each month during the six months. Through an action planning and implementation process, care communities are guided to make organization-wide, measurable changes in the areas of (1) policies and procedures, (2) education and training, and/or (3) care practices to increase and maintain person-centered care practices as outlined in the DCPR. Coaches provide ongoing support to the care community through telephone and email support between meetings. Control group will not receive any coaching intervention but receive monthly email (e.g., newsletter about Alzheimer's Association but not related to outcomes) from coaches for check-in. Alzheimer's Association (AA) hires coaches in study areas based on their skills, experiences, interests and enthusiasm. Each coach identifies and invites long-term care (i.e., nursing home and assisted living) communities using existing relationships between the AA Chapter and those communities. In addition, AA staff will work with a national and/or state-wide networking group /association, as well as the Association's Dementia Care Provider Round Tables. The investigators will also pull the list of nursing homes in the study areas from publicly available data (e.g., Definitive Healthcare). Once each care community is selected and has agreed to participate, DCPR coaches will request that the care community identify 4-6 staff members to serve on a Care Team. The consented care communities are randomly assigned to either a control or intervention group (1: 1 block randomization).

ELIGIBILITY:
Inclusion Criteria:

* Licensed skilled nursing facilities
* Licensed assisted living facilities
* Located in the state of Ohio

Exclusion Criteria:

* Under the age of 18
* Without documented endorsement for participation from facility leadership

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
Employee Satisfaction | pre, immediately post, and 3-month post
  Employee satisfaction was measured using the Centers for Medicare & Medicaid Services (CMS)'s Nursing Home Employee Satisfaction Survey. This tool contains 5 topic areas, including job satisfaction (9 items), team building and communication (10 items), scheduling and staffing (4 items), training (6 items), and management and leadership (6 items). Participants will answer on a scale from 1 (strongly disagree) to 5 (strongly agree). Average score overall and by topic areas will be calculated (range = 1 - 5), where a higher score indicates greater employee satisfaction.

SECONDARY OUTCOMES:
Dementia care confidence | pre, immediately post, and 3-month post
  Dementia care confidence is measured using the Confidence in Dementia Scale (CODES) The nine-item self-report questionnaire is scored on a 5-point scale with anchored ratings of 'not able', 'slightly able', 'somewhat able', 'mostly able', 'very able'. Total score ranges from 9 to 45, with a higher score signifying better confidence in working with people with dementia.
Person-centered practices | pre, immediately post, and 3-month post.
  Person-centered practices are measured using the Toolkit for Person-Centeredness in Assisted Living (workplace practices, individualized care and services, and caregiver-resident relationships domains). From this tool, three areas will be measured, including workplace practices (23 items), individualized care and services (8 items), and caregiver-resident relationships domains (7 items). Participants will answer on a 5-point scale from 1 (strongly disagree) to 5 (strongly agree). Average score overall and by areas will be calculated, and then multiply the average scores by 25. Total scores overall and by areas range between 25 and 100, with a higher score representing more person-centeredness.

OTHER OUTCOMES:
Staff Turnover | Monthly, from the month pre-intervention to 3 months after completion of the intervention (9 times)
  Turnover rates are assessed monthly from pre-intervention to 3 months after completion of the intervention (9 times) for direct care staff (i.e., certified nursing assistants (CNAs), care aids and other equivalent, front-line care staff), health and social services staff (i.e., registered nurses (RNs), licensed practical nurses (LPNs), social services, activities staff), and leadership staff (i.e., directors of nursing, unit leaders, licensed administrators). Turnover rates (%) are calculated using the National Nursing Home Quality Improvement Campaign Staff Stability Tracking Tool v2.2, dividing the number terminated as of the last day of the month by the number employed as of the first day of the month.

CONTACTS AND LOCATIONS:
Overall Officials: Sam Fazio, PhD, Principal Investigator — Alzheimer's Association
Locations (1):
- Alzheimer's Association, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fazio S, Pace D, Maslow K, Zimmerman S, Kallmyer B. Alzheimer's Association Dementia Care Practice Recommendations. Gerontologist. 2018 Jan 18;58(suppl_1):S1-S9. doi: 10.1093/geront/gnx182. No abstract available. PMID 29361074